CLINICAL TRIAL: NCT03149068
Title: Studying the Relationship Between Mean Platelet Volume and Neutrophil/ Lymphocyte Ratio With Inflammation and Proteinuria in Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, walaa soliman, assuit, Assiut University
Other Study IDs: Assuit University 96
Record Dates: First submitted 2017-05-02; First posted 2017-05-11 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Evaluation of Early Inflammatory Process in CKD

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 75 patient: Seventy five (75) CKD patients in different stages will be included in our study from Nephrology unit, Internal Medicine department, Assuit University Hospital
- 25 healthy control: twenty five (25) age and sex matched apparently healthy individuals will be enrolled as controls

SUMMARY:
Inflammation begins during early stages of CKD in which neutrophil counts are increased, whereas lymphocyte counts are decreased during inflammation. In addition to known conventional indications of inflammation such as C-reactive protein (CRP), fibrinogen, erythrocyte sedimentation rate, several interleukins and tumor necrotizing factor alpha, Neutrophil-to-lymphocyte ratio (NLR) has increasingly been reported as a measure of systemic inflammation (Okyay G U et al 2013 and Yilmaz G et al ,2017) Several recent studies have shown that mean platelet volume (MPV) is also increased during inflammation and may be associated with poorer prognosis in CKD (Yilmaz G et al ,2017).

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a worldwide problem and its incidence is steadily increasing. Kidney Disease Outcomes Quality Initiative (K/DOQI) of the National Kidney Foundation (NKF) defines chronic kidney disease as either kidney damage or a decreased kidney glomerular filtration rate (GFR) of less than 60 mL/min/1.73 m2 for 3 or more months (Levey AS.,2011). Whatever the underlying etiology, the destruction of renal mass with irreversible sclerosis and loss of nephrons leads to a progressive decline in GFR. CKD progression is associated with high morbidity and mortality (Sanz AB.,2014) .The early detection of CKD is important and early treatment may reduce adverse outcomes associated with CKD and slow or even prevent the progression of the disease. Therefore, the detection of CKD at early stages is an important public health issue (Katherine T.,2015).

Cardiovascular disease is a leading cause of death in patients with chronic kidney disease (CKD), for whom the cardiovascular mortality rate is 15 to 30 times higher than in the general population. The underlying pathological state is caused by a complex interplay of traditional and nontraditional risk factors that results in atherosclerosis, arteriosclerosis, and altered cardiac morphological characteristics. (Effat et al 2012) Several factors are associated with the onset and progression of CKD, such as obesity, hypertension and diabetes mellitus. Beyond these factors, there is evidence of a pathophysiological role for inflammation in CKD. Inflammation actively participates in the mechanisms of renal damage progression in diseases of several etiologies (Akchurin OM and Kaskel F, 2015). In glomerular diseases, for example, the following sequence is believed to occur: 1) persistent glomerular injury produces capillary hypertension, with increased glomerular filtration and passage of proteins into the tubular fluid; 2) glomerular proteinuria increases the production of angiotensin II and promotes liberation of inflammatory mediators (cytokines and chemokines), which induce the renal interstitial build-up of mononuclear cells; 3) the initial neutrophil recruiting is replaced by macrophages and T lymphocytes, which unleash the immune response producing interstitial nephritis; 4) tubular cells respond to this inflammatory process with injury to their basement membrane and with the epithelial-mesenchymal transition, becoming interstitial fibroblasts; 5) The formed fibroblasts produce collagen which, in turn, injuries the renal vessels and tubules, eventually generating a cellular scar (Vianna H R et al 2011).

Inflammation begins during early stages of CKD in which neutrophil counts are increased, whereas lymphocyte counts are decreased during inflammation. In addition to known conventional indications of inflammation such as C-reactive protein (CRP), fibrinogen, erythrocyte sedimentation rate, several interleukins and tumor necrotizing factor alpha, Neutrophil-to-lymphocyte ratio (NLR) has increasingly been reported as a measure of systemic inflammation (Okyay G U et al 2013 and Yilmaz G et al ,2017) . It is a simple parameter to assess easily the inflammatory status of a subject and has proven its usefulness in the stratification of mortality in major cardiac events, as a strong prognostic factor in several types of cancers , or as a predictor and a marker of inflammatory or infectious pathologies (ex., pediatric appendicitis) and postoperative complications (Forget P et al 2017). Recent studies have emphasized that NLR could be used as an indication for inflammation and may be associated with poorer prognosis in CKD (Yilmaz G et al ,2017) .

Several recent studies have shown that mean platelet volume (MPV) is also increased during inflammation and may be associated with poorer prognosis in CKD (Yilmaz G et al ,2017). Platelet activation in patients with chronic kidney disease (CKD) may contribute to cardiovascular mortality. The relationship between mean platelet volume (MPV) and coronary artery disease, atherosclerotic vascular pathologies, and platelet aggregation in CKD is not well established (Altun E et al 2016).

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for participation in the study if :

  1. Patients between the ages of 19-65 years
  2. CKD patient in stages 2,3,4
  3. GFR values of 15-89 mL/min/1.73 m2
  4. Body mass index ( BMI ) <35 kg/ m2

Exclusion Criteria:

* Patients were excluded from the study if :

  1. Diabetes Mellitus patients,
  2. Patients with any active infection,
  3. Patients with any malignancy,
  4. Patients with coronary artery disease ,
  5. Patients on steroids and , or immunosuppressive drugs

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Patients will be subjected to the following:
  1.A full history and thorough clinical evaluation. 2. Estimated GFR of patients will calculated using CKD-epidemiology collaboration formula, Modified Medried formula: (Coresh J .,2007). 3.Biochemistry and hemograms will be done for all patients and controls: i. peripheral blood count :
  * The neutrophil to lymphocyte ratio (NLR) will be calculated. NLR values are normal ,if the value is between 0.78 and 3.58.( Forget P et al 2017).
  * Mean platelet volume (MPV) : 7.2-11.7 fL (Hilmi Demiri et al 2011) Then, the relationship between MPV/NLR will be evaluated ii. urine analysis . iii. renal function tests iv. 24 hour urine protein if proteinuria is detected v. 24 hour urine microalbumin vi. liver function tests vii. lipid profile after fasting 12 hours viii. serum uric acid ix. CRP x.serum fibrinogen level
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-07-01 (Estimated); Primary Completion 2018-05-01 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
Studying the Relationship Between Mean Platelet Volume and Neutrophil/ Lymphocyte Ratio With Inflammation and Proteinuria in Chronic Kidney Disease | one year
  The relationship between (MPV) and (NLR) with inflammation and proteinuria in patients with CKD at stage 2 , 3 and 4 by simple parameters.

IPD SHARING:
Plan to Share IPD: Undecided